CLINICAL TRIAL: NCT07395401
Title: Clinical and Radiographic Evaluation of Zinc Oxide Eugenol (ZOE) and Iodoform-Calcium Hydroxide (Metapex) as Filling Materials in Primary Molar Root Canals Prepared by Rotary and Manual Files: (Randomized Control Trial Study)
Brief Title: Evaluation of Zinc Oxide Eugenol and Iodoform-Calcium Hydroxide as Filling Materials in Primary Molar Root Canals Prepared by Rotary and Manual Files
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Nanis Nasser Anwar Moustafa, teacher assistant at pediatric dentistry department, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U MSA Nanis
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Carious Primary Molars Indicated for Pulpectomy
Keywords: Iodoform-Calcium Hydroxide; Metapex; Zinc Oxide Eugenol; Manual Instrumentation Method; Rotary Instrumentation Method; pulpectomy; primary molars; radiographic assessment; clinical assessment
MeSH Terms: interventions — Metapex; Zinc Oxide-Eugenol Cement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A: Manual Instrumentation and Metapex (Experimental): Primary molar teeth will undergo pulpectomy using Manual instrumentation followed by obturation with iodoform-calcium hydroxide paste (Metapex).
  Interventions: Procedure: Manual Instrumentation; Drug: Iodoform-Calcium Hydroxide (Metapex)
- Arm B: Rotary Instrumentation and Metapex (Experimental): Primary molar teeth will undergo pulpectomy using rotary instrumentation followed by obturation with iodoform-calcium hydroxide paste (Metapex).
  Interventions: Drug: Iodoform-Calcium Hydroxide (Metapex); Procedure: Rotary Instrumentation
- Arm C: Manual Instrumentation and ZOE (Active Comparator): Primary molar teeth will undergo pulpectomy using manual instrumentation followed by obturation with zinc oxide eugenol (ZOE).
  Interventions: Procedure: Manual Instrumentation; Drug: Zinc Oxide Eugenol (ZOE)
- Arm D: Rotary Instrumentation and ZOE (Active Comparator): Primary molar teeth will undergo pulpectomy using rotary instrumentation followed by obturation with zinc oxide eugenol (ZOE).
  Interventions: Procedure: Rotary Instrumentation; Drug: Zinc Oxide Eugenol (ZOE)

INTERVENTIONS:
Procedure: Manual Instrumentation — Root canal preparation of primary molars will be performed using manual stainless-steel hand files with conventional step-back technique for cleaning and shaping of the root canals.
  Arms: Arm A: Manual Instrumentation and Metapex; Arm C: Manual Instrumentation and ZOE
Drug: Iodoform-Calcium Hydroxide (Metapex) — Metapex (iodoform-calcium hydroxide paste) will be used as the obturating material for filling the prepared root canals of primary molars following pulpectomy.
  Arms: Arm A: Manual Instrumentation and Metapex; Arm B: Rotary Instrumentation and Metapex
Procedure: Rotary Instrumentation — Root canal preparation of primary molars will be performed using nickel-titanium rotary instruments according to the manufacturer's instructions to achieve effective cleaning and shaping of the root canals.
  Arms: Arm B: Rotary Instrumentation and Metapex; Arm D: Rotary Instrumentation and ZOE
Drug: Zinc Oxide Eugenol (ZOE) — Zinc oxide eugenol paste will be used as the obturating material for filling the prepared root canals of primary molars following pulpectomy.
  Arms: Arm C: Manual Instrumentation and ZOE; Arm D: Rotary Instrumentation and ZOE

SUMMARY:
This randomized controlled clinical trial aims to compare the clinical and radiographic outcomes of Zinc Oxide Eugenol (ZOE) and Iodoform-Calcium Hydroxide (Metapex) as root canal filling materials in primary molars prepared using either rotary or manual instrumentation techniques. Forty-four teeth from children aged 5-8 years indicated for pulpectomy will be randomly allocated into four equal groups based on the combination of instrumentation method and filling material. Clinical parameters-pain, mobility, and sensitivity-will be assessed using standardized scales, while radiographic outcomes, including root resorption and bone density, will be evaluated using Cone Beam Computed Tomography (CBCT) at baseline, 6 months, and 12 months. The study seeks to determine which obturation material and canal preparation technique yield superior healing, adaptation, and resorption compatible with the physiological process of primary tooth exfoliation. Findings are expected to inform evidence-based selection of endodontic materials and instrumentation methods in pediatric dentistry.

DETAILED DESCRIPTION:
Preservation of primary teeth is essential for maintaining proper mastication, speech development, and arch integrity, as well as for preventing psychological and functional complications arising from premature tooth loss. Pulpectomy remains the treatment of choice for irreversibly infected or necrotic primary teeth, yet the complex root canal morphology, resorptive nature of primary roots, and behavioral management challenges make such procedures technically demanding.

An ideal root canal filling material for primary teeth should be antibacterial, biocompatible, radiopaque, and resorbable at a rate consistent with natural root resorption. It must also be easily manipulated, removable if necessary, and capable of hermetic sealing. Among the commonly used materials, Zinc Oxide Eugenol (ZOE) has long been considered the standard due to its antimicrobial and sealing properties; however, its slow resorption and potential for periapical irritation are significant drawbacks. Conversely, Metapex, a premixed iodoform-calcium hydroxide paste, exhibits superior biocompatibility, antibacterial effects, and resorption rates that align more closely with physiological root resorption, making it a promising alternative.

Similarly, biomechanical preparation of root canals can be performed manually or using nickel-titanium (NiTi) rotary systems. Manual instrumentation provides tactile feedback and precision but is time-consuming and operator-dependent. Rotary systems, on the other hand, offer improved efficiency, shaping consistency, and reduced chair time-important factors in managing pediatric patients-though they require training and careful use to prevent over-preparation.

This study will enroll 44 primary molars from cooperative, systemically healthy children aged 5-8 years who are indicated for pulpectomy. The teeth will be randomly allocated into four groups:

Rotary instrumentation with Metapex,

Rotary instrumentation with ZOE,

Manual instrumentation with Metapex, and

Manual instrumentation with ZOE.

Clinical evaluation will include assessment of pain using the Wong-Baker FACES Pain Rating Scale, mobility using Miller's Mobility Index, and sensitivity using the Numeric Rating Scale (NRS). Radiographic evaluation will be performed using CBCT at baseline, 6, and 12 months to assess root resorption and bone density changes. The primary outcome is radiographic success, defined by physiological resorption and bone healing, while secondary outcomes include clinical success indicators such as absence of pain, swelling, or abnormal mobility.

Data will be statistically analyzed using SPSS (v24). Quantitative variables will be tested for normality and compared using ANOVA or Kruskal-Wallis tests, while qualitative data will be analyzed using Chi-square tests.

The findings are expected to clarify whether Metapex or ZOE, when used with rotary or manual preparation techniques, provides superior clinical and radiographic outcomes. Ultimately, the results may guide clinicians toward more effective, biocompatible, and time-efficient pulpectomy protocols in pediatric endodontics, contributing to improved long-term oral health outcomes in children.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy cooperative children indicated for partial pulpectomy.
2. Restorable primary molars.
3. No mobility, or external pathological root resorption.

Exclusion Criteria:

1. Uncooperative children.
2. Children with systemic medical illness.
3. More than 2/3 of root resorbed.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success | Baseline, 6 months, and 12 months
  Radiographic success will be assessed by evaluating root resorption in treated primary molars. Cone Beam Computed Tomography (CBCT) will be used to measure the degree of root resorption in millimeters, allowing comparison between zinc oxide eugenol (ZOE) and iodoform-calcium hydroxide (Metapex) obturation materials in canals prepared by rotary and manual instrumentation techniques.

SECONDARY OUTCOMES:
Postoperative Pain | Baseline, 6 months, and 12 months
  Pain will be evaluated using the Wong-Baker FACES Pain Rating Scale. Patients will self-report pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable) during follow-up visits after pulpectomy.
Tooth Mobility | Baseline, 6 months, and 12 months
  Tooth mobility will be assessed clinically using Miller's Mobility Index by applying gentle pressure with a dental instrument to evaluate the degree of horizontal and vertical movement of the treated primary molars where 0 (no mobility) to 3 (more than 1mm vertical and horizontal mobility) during clinical examination.
Tooth Sensitivity | Baseline, 6 months, and 12 months
  Tooth sensitivity will be evaluated using the Numeric Rating Scale (NRS), where patients will rate sensitivity from 0 (no sensitivity) to 10 (extreme sensitivity) during clinical examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, MSA University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No